CLINICAL TRIAL: NCT05287321
Title: The Efficacy of Aspirin Combined With Hydroxychloroquine Treatment in High Risk Pregnancies for Preeclampsia: a Multicenter, Open-label, Single Arm Trial, Investigator Initiated Study
Brief Title: The Efficacy of Aspirin Combined With Hydroxychloroquine Treatment in High Risk Pregnancies for Preeclampsia
Acronym: HUGS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yoo-min Kim (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor-Investigator, Yoo-min Kim, Assistant professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Organization: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2112-014-487
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aspirin 100mg + Hydroxychloroquine 200mg (Experimental): Aspirin 100mg 1T daily PO + Hydroxychloroquine 200mg 1T daily PO
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 200mg with Aspirin 100mg
  Other Names: Plaquenil

SUMMARY:
This study is prospective, single arm group ,open label, and multicenter trial (with two parallel-group [Hydroxychloroquine 200mg with Aspirin 100mg or Aspirin 100mg])

DETAILED DESCRIPTION:
This study is prospective, open label, and multicenter trial [Hydroxychloroquine 200mg with Aspirin 100mg]

The study population consists of the singleton pregnancy at high risk for preeclampsia who had adverse pregnancy outcome (preeclampsia or fetal growth restriction or intrauterine fetal death) in previous pregnancy.

After randomisation, participants are assigned to receive hydroxychloroquine 200mg with aspirin 100mg per day or aspirin 100mg per day. Treatment is initiated between 12 and 22 weeks' gestation and stopped at 36 weeks' gestation.

The medication adherence to dosing should be maintained at more than 80%.

ELIGIBILITY:
Inclusion Criteria:

1. The singleton pregnant women aged from 19 to 50 years
2. Includes at least one factors of the below

   ① History of preeclampsia

   ② History of fetal growth restriction

   ③ History of intrauterine fetal death
3. Women who have agreed to enroll in the study and given their informed consent

Exclusion Criteria:

1. Indication to a treatment according to the severe cardiovascular, immune, respiratory, gastrointestinal/liver and biliary system, kidney and urinary system, nervous system, musculoskeletal system, psychiatric, infectious disease and malignancy (However, the participation of the trial is allowed by the investigator based on medically necessary.)
2. Previous inclusion in other intervention study within 3 months of screening (except for non-interventional observational studies)
3. Major malformation of the fetus is diagnosed at 11-13 weeks of gestation
4. Elevated blood concentrations of creatinine more than double the normal value
5. Elevated blood concentrations of liver transaminases (AST(GOT) or ALT(GPT)) more than three times the normal value
6. Conditions related with aspirin treatment

   * Previous exposure within 28 days of screening
   * Previous NSAID exposure within 28 days of screening
   * Bleeding disorder (von Willebrand's disease, peptic ulceration)
   * Hypersensitivity to aspirin
7. Conditions related with hydroxychloroquine treatment

   * Previous exposure within 28 days of screening
   * Hypersensitivity to hydroxychloroquine and 4-aminoquinoline compounds
   * Maculopathy
   * Medications that has potential for visual disturbance
   * Women who have potential for changes in the retina or visual impairment by 4-aminoquinoline compounds
   * Galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
   * Prolonged QT interval on EKG (congenital or acquired) or The risk factors of QT prolongation (heart failure, arrhythmia, myocardial ischemia)
   * Low level of potassium in the blood
   * Low level of magnesium in the blood
8. Not suitable for participant based on medical evidence by investigator

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite morbidity | gestational period
  Preeclampsia, Fetal growth restriction, Intrauterine fetal death, preterm delviery (<37weeks)

SECONDARY OUTCOMES:
Severe preeclampsia | gestational period
  with severe features: severe features are uncontrolled BP (systolic BP > 160mm Hg or diastolic BP > 110mm Hg on two occasions at least 4hours apart), persistent epigastric pain, new onset headaches, pulmonary edema, thrombocytopenia (platelet count <100,000/µL), elevated liver enzymes (at twice the upper limit), impaired renal insufficiency (serum creatinine > 1.1mg/dL)
early preterm birth | gestational period
  between 23+0wks and 33+6weeks
Late preterm birth | gestational period
  delivery between 34+0 to 36+6 weeks
Severe Fetal growh restrection | gestational period
  <3% and <5% for a given gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-min Kim, MD, Principal Investigator — Chung-Ang University Gwangmyeong Hospital
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YM, Seong J, Kim JH, Nam G, Kim GJ, Cha HH, Seong WJ, Sung JH, Choi SJ, Oh SY, Roh CR. Efficacy of combining aspirin with hydroxychloroquine in pregnancies at high risk for pre-eclampsia: a prospective, multicentre, open-label, single-arm clinical trial, investigator-initiated study (HUGS study). BMJ Open. 2024 Dec 10;14(12):e081610. doi: 10.1136/bmjopen-2023-081610. PMID 39658277